CLINICAL TRIAL: NCT03279159
Title: Hydrating Efficacy and Tolerance Evaluation of a Face Cream
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Dermatologist, Principal Investigator, Derming SRL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E0617
Record Dates: First submitted 2017-09-04; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-06

CONDITIONS: Dry and Damaged Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jaluronius CS cream (Difa Cooper S.p.a, Italy) (Experimental)
  Interventions: Other: Jaluronius CS cream short term evaluation; Other: Jaluronius CS cream long term evaluation

INTERVENTIONS:
Other: Jaluronius CS cream short term evaluation — Short term evaluation to investigate the hydrating activity of a single application of the study product on the forearms (volar surface) after repeated stripping procedure,measured immediately after stripping execution (T0i), 1,8 and 24 hour/s after product application (T1h, T8h and T24h).
Other: Jaluronius CS cream long term evaluation — Long term evaluation to investigate the hydrating activity of the repeated application of the study product on the face (twice a day, for an uninterrupted period of 8 weeks), measured at basal visit (T0) and after 4 and 8 week-treatment (T4, T8)

SUMMARY:
Aim of the study was to evaluate by non-invasive instrumental evaluations tolerance and hydrating activity of a face topic product, to be applied twice a day, morning and evening, for an uninterrupted period of 8 weeks, by volunteers of both sexes, aged 45-60, who meet the inclusion and exclusion criteria required by the study procedure .

It was also aim of this study to evaluate the hydrating activity of a single product application on the skin damaged by repeated stripping corneum (short term evaluation versus untreated control area).

ELIGIBILITY:
Inclusion Criteria:

* both sexes,
* age 45-60 years,
* caucasian subjects,
* agreeing to present at each study visit without make-up,
* accepting to follow the instructions received by the investigator,
* accepting to not change their habits regarding food, physical activity, face cleansing and make- up use,
* agreeing not to apply or take any product or use face massages or other means known to improve skin wrinkle and skin qualities during the entire duration of the study,
* accepting not to expose their face to strong UV irradiation (UV session, or sun bathes), during the entire duration of the study,
* no participation in a similar study currently or during the previous 3 months
* accepting to sign the Informed consent form.

Exclusion Criteria:

* Pregnancy (only for female subjects),
* lactation (only for female subjects),
* sensitivity to the test product or its ingredients (to be assessed by the investigator during the baseline visit),
* subjects whose insufficient adhesion to the study protocol is foreseeable.
* presence of cutaneous disease on the tested area as lesions, scars, malformations,
* recurrent facial/labial herpes,
* clinical and significant skin condition on the test area (e.g. active eczema, dermatitis, psoriasis etc.).
* endocrine disease,
* hepatic disorder,
* renal disorder,
* cardiac disorder,
* pulmonary disease,
* cancer,
* neurological or psychological disease,
* inflammatory/immunosuppressive disease,
* drug allergy.
* anti-inflammatory drugs, anti-histaminic, topic (application on the face) and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of hormonal treatment starting more than 1 year ago),
* using of drugs or dietary supplements able to influence the test results in the investigator opinion.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Change of superficial skin hydration after a single product application | Immediately after stripping (T0i), 1 hour after product application (T1h), 8 hours after product application (T8h), 24 hours after product application (T24h)
  Variation of skin electrical capacitance value measured with Corneometer CM825 (Courage - Khazaka, Köln, Germany) after a single product application on the skin area damaged by corneum stripping
Change of transepidermal water loss (TEWL) after a single product application | Immediately after stripping (T0i), 1 hour after product application (T1h), 8 hours after product application (T8h), 24 hours after product application (T24h)
  Variation of transepidermal water loss value measured with Tewameter® TM300 (MPA 5 Courage-Khazaka, Germany) after a single product application on the skin area damaged by corneum stripping
Change of superficial skin hydration after repeated product application | Baseline (T0), 4 weeks (T4), 8 weeks (T8)
  Variation of skin electrical capacitance value measured with Corneometer CM825 (Courage - Khazaka, Köln, Germany) after repeated product application on the face
Change of deep skin hydration after repeated product application | Baseline (T0), 4 weeks (T4), 8 weeks (T8)
  Variation of tissue dielectric constant value of deep skin layers measured with MoistureMeterD (Delfin Technologies, Kuopio - Finland) after repeated product application on the face

CONTACTS AND LOCATIONS:
Locations (1):
- DERMING, Monza, Monza-brianza, Italy